CLINICAL TRIAL: NCT04963543
Title: Evaluation of Comfort in Symptomatic Contact Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DEJ475-E003
Record Dates: First submitted 2021-07-06; First posted 2021-07-15 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: Ocular Comfort
Keywords: Contact Lenses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FID123238 (Experimental): FID123238 applied to the ocular surface, 1 application per day, for five consecutive days
  Interventions: Other: FID123238

INTERVENTIONS:
Other: FID123238 — Lubricant applied to the ocular surface

SUMMARY:
The purpose of this study is to evaluate the comfort of an ocular lubricant in symptomatic contact lens wearers. This study will be conducted in Canada.

DETAILED DESCRIPTION:
The duration of individual participation is six days.

ELIGIBILITY:
Key Inclusion Criteria:

* Is able to understand and sign an approved information consent letter;
* Habitually wears daily disposable soft contact lenses in both eyes;
* Is able to achieve 20/40 or better monocular VA with habitual contact lenses;
* Has a pair of spectacles for vision correction.
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Routinely sleeps in habitual contact lenses;
* Has any known active ocular disease and/or infection;
* Is pregnant or lactating;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
Comfort, collected for each eye | Up to Day 6
  A visual analogue scale will be used

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Dry Eye, Study Director — Alcon Research, LLC
Locations (1):
- Alcon Investigative Site 6189, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No